CLINICAL TRIAL: NCT04292119
Title: A Phase IB/II Study of Lorlatinib Combinations in Anaplastic Lymphoma Kinase-Rearranged Lung Cancer
Brief Title: Lorlatinib Combinations in Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Array BioPharma (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Ibiayi Dagogo-Jack, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-629
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Anaplastic Lymphoma Kinase Gene Translocation; ROS1 Rearrangement; Relapsed Cancer; MET Amplification; Resistant Cancer; NSCLC
Keywords: Lung Cancer; Anaplastic Lymphoma Kinase Rearrangement; ROS1 Rearrangement; Relapsed Cancer; Resistant Cancer; MET Amplification; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Recurrence | interventions — lorlatinib; Crizotinib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lorlatinib and Crizotinib (Experimental): * The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits.
  * Phase 1 (the dose-finding portion of the study) will follow a standard 3+3 design. Enrollment to the different study arms will occur in parallel.
    * Lorlatinib will be administered orally once daily at a predetermined dose for 28 days
    * Crizotinib will be administered orally twice daily at a predetermined dose for 28 days
  * Phase II patients will be treated with Lorlatinib and Crizotinib at a dose recommended based on the phase I study.
  Interventions: Drug: Lorlatinib; Drug: Crizotinib
- Lorlatinib and Binimetinib (Experimental): * The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits.
  * The phase I part of the study will follow a standard 3+3 design. Enrollment to the different study arms will occur in parallel.
    * Lorlatinib will be administered orally once daily at a predetermined dose for 28 days
    * Binimetinib will be administered orally twice daily at a predetermined dose for 28 days.
  * Phase II patients will be treated with Lorlatinib + Binimetinib at a dose recommended based on the phase I study.
  Interventions: Drug: Lorlatinib; Drug: Binimetinib
- Lorlatinib and TNO155 (Experimental): * The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits.
  * The phase I part of the study will follow a standard 3+3 design. Enrollment to the different study arms will occur in parallel.
    * Lorlatinib will be administered orally once daily at a predetermined dose for 21 days
    * TNO155 will be administered orally once daily at a predetermined dose for 14 out of 21 days.
  * Phase II patients will be treated with Lorlatinib + TNO155 at a dose recommended based on the phase I study.
  Interventions: Drug: Lorlatinib; Drug: TNO155

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib will be taken orally once daily for 28 days when combined with crizotinib or binimetinib. Lorlatinib will be taken orally once daily for 21 days when combined with TNO155.
  Crizotinib taken orally twice daily for 28 days.
  Other Names: Lorbrena
Drug: Crizotinib — Crizotinib will be taken orally twice daily for 28 days.
  Binimetnib taken orally twice daily for 28 days.
  Other Names: Xalkori
  Arms: Lorlatinib and Crizotinib
Drug: Binimetinib — Binimetinib will be taken orally twice daily for 28 days.
  Other Names: Mektovi
  Arms: Lorlatinib and Binimetinib
Drug: TNO155 — TNO155 will be taken orally once daily for 14 days.
  Arms: Lorlatinib and TNO155

SUMMARY:
This research study is evaluating Lorlatinib in combination with Crizotinib, Binimetinib, or TNO155 as a possible treatment for either anaplastic lymphoma kinase (ALK)-positive lung cancer or ROS1-positive lung cancer.

* This research study involves four study drugs.
* Lorlatinib
* Binimetinib
* Crizotinib
* TNO155

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial of three investigational combinations for treatment of either anaplastic lymphoma kinase (ALK)-positive or ROS1-positive lung cancer. The three drug combinations being tested are (1) Lorlatinib combined with Crizotinib and (2) Lorlatinib combined with Binimetinib and (3) Lorlatinib combined with TNO155.

* Lorlatinib is an oral ALK and ROS1 inhibitor. The US Food and Drug Administration (FDA) has approved Lorlatinib for treatment of ALK-positive lung cancer. The FDA has not approved Lorlatinib for treatment of ROS1-positive lung cancer.
* Crizotinib is an oral ALK and MET inhibitor. The FDA has approved Crizotinib for treatment of ALK-positive lung cancer. Crizotinib is not approved by the FDA for the treatment of MET-positive lung cancer. This study will test crizotinib's ability to block MET signaling. Crizotinib is not approved by the FDA for treatment of ROS1-positive lung cancer.
* Binimetinib is an oral MEK inhibitor. The FDA has not approved binimetinib for treatment of ALK-positive or ROS1-positive lung cancer but it has been approved for other uses.
* TNO155 is an oral SHP2 inhibitor. The FDA has not approved TNO155 for the treatment of any disease, including ALK-positive or ROS1-positive lung cancer. It is an investigational drug.
* The FDA has not approved the combination of Lorlatinib with Binimetinib, Crizotinib, or TNO155 as a treatment for any disease.

The research study procedures include screening for eligibility and study treatment which will include evaluations and follow up visits.

* Patients will undergo screening and those who fulfill the eligibility criteria will be assigned to receive either the combination of Lorlatinib and Crizotinib, the combination of Lorlatinib and Binimetinib, or the combination of Lorlatinib and TNO155. Patients with ALK-positive or ROS1-positive lung cancer who have extra copies of the MET growth signal (MET amplification) will be assigned to receive the Lorlatinib and Crizotinib combination. All other patients will be randomly assigned to receive one of the combinations.
* This study consists of 2 parts:

  * Phase I:

    * The investigators are looking to determine whether combining Lorlatinib with either Binimetinib, Crizotinib, or TNO155 is well tolerated and to understand how treatment with the two drugs affects cancer cells and impacts growth signals.
    * Not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
  * Phase II:

    * The Phase II study will test the safest doses of the combinations (as established in the Phase I study) in a larger group of patients.
    * It is expected that about 96 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years.
* Histologically or cytologically confirmed diagnosis of metastatic non-small cell lung cancer (Stage IV, AJCC v7.0) that carries an ALK or ROS1 rearrangement (ROS1-positive patients will only be allowed in dose escalation) as determined using a local diagnostic test or a commercial test or by the Food and Drug Administration (FDA)-approved FISH test, using Vysis® ALK Break apart FISH Probe, or the Ventana® immunohistochemistry (IHC) test.
* Disease progression or intolerance to at least one tyrosine kinase inhibitor
* At least one measurable lesion as defined by RECIST version 1.1. Previously irradiated lesions are not measurable unless the lesion has demonstrated clear progression after radiation.
* ECOG performance status ≤ 2
* Life expectancy of greater than 12 weeks
* Patients must be willing to undergo serial biopsies and have disease accessible to pretreatment biopsy. A cell block from a pleural effusion or ascites may be substituted for a core biopsy. In select cases, patients may be allowed to enroll without a pre-treatment biopsy and/or continue treatment without an on-treatment biopsy after speaking with the Overall Principal Investigator if performing the biopsy is technically challenging, poses significant risk to the patient, or may result in significant discomfort. If a pre-treatment biopsy is not performed, archival tissue will be used for correlative studies, specifically plasma-tissue comparisons.
* Able to swallow and retain orally administered medication. Does not have any clinically significant gastrointestinal abnormalities, such as malabsorption syndrome or major resection of the stomach or small bowel that may alter absorption of the medication.
* A minimum washout period of 5 days or 5 half-lives between the last dose of tyrosine kinase inhibitor therapy and the first dose of study treatment is required (whichever is shorter). A shorter washout period may be considered in the event of disease flare, after discussion with the Overall Principal Investigator. No washout is required if the most recent anti-neoplastic therapy is lorlatinib.
* Patients must have recovered from treatment toxicities to ≤ Grade 1 or to their pretreatment levels except for adverse events that in the investigator's judgment do not constitute a safety risk for the patient.
* Patients can either be chemotherapy-naive or have received chemotherapy for locally-advanced or metastatic disease. Acute effects of therapy must have resolved to baseline severity or to CTCAE grade ≤1 except for adverse events that in the investigator's judgment do not constitute a safety risk for the patient.
* Recovery from effects of any major surgery or significant traumatic injury at least 28 days before the first dose of study treatment.
* For all women of childbearing potential, a negative pregnancy test must be obtained at the baseline visit before starting study treatment. For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 90 days after the last dose of study drug.

  * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide.
* For men: agreement to remain abstinent or use a barrier method of contraception (e.g., condom) during the treatment period and for at least 90 days after the last dose of study drug and agreement to refrain from donating sperm during this same period
* Men with a pregnant partner must agree to remain abstinent or use a condom for the duration of the pregnancy.
* Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Patients with untreated, controlled asymptomatic CNS lesions are permitted to enroll aslong as the CNS was not a site of progressive disease on lorlatinib monotherapy. If the CNS was a site of progressive disease on lorlatinib monotherapy, treatment of CNS lesions is required for enrollment. If CNS lesions are resected, a washout period of at least 28 days is required. This period may be shortened to 14 days with Overall PI approval.
* The use of seizure prophylaxis is allowed as long as patients are taking non-enzyme inducing anti-epileptic drugs (non-EIAED). If patients were previously on EIAEDs and these have been discontinued, they must have been discontinued for at least 7 days prior to treatment start. If patients require an anti-epileptic medication, then a CYP3A4 non-EIAED can be used such as levetiracetam, valproic acid, gabapentin, topiramate or lacosamide.
* Patients requiring steroids for control of CNS metastases must be at a stable or decreasing dose for at least 1 week prior to enrollment
* Patients with asymptomatic leptomeningeal disease are eligible for participation in this trial. However, patients who had progression of leptomeningeal disease on lorlatinib will be required to undergo CNS radiation to meet eligibility.

Exclusion Criteria:

* Participants who have had chemotherapy or immunotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Participation in other studies involving investigational drug(s) within 1 week prior to study entry and/or during study participation. If the half-life of the investigational drug is known, then a period of 5 half-lives is required (or 1 week whichever is shorter) is required between discontinuing the investigational drug and starting study treatment.
* Radiation therapy (except palliative to relieve bone pain) within 7 days of study entry. Palliative radiation (≤ 10 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have been completed at least 48 hours prior to study entry. Whole brain radiation and radiation for leptomeningeal metastasis must have been completed at least 7 days prior to study entry. Acute effects of radiation must have resolved to baseline severity or to CTCAE grade ≤1 except for adverse events that in the investigator's judgment do not constitute a safety risk for the patient.
* Pregnant or lactating women.
* Patients with predisposing characteristics for acute pancreatitis per the investigator's judgment (e.g. uncontrolled hyperglycemia, current symptomatic gallstone disease) in the 2 weeks prior to randomization
* History of hypersensitivity to lorlatinib or any of its excipients. In addition, subjects who are unable to tolerate the 50 mg dose of lorlatinib will not be permitted to enroll unless doses of lorlatinib below the entry level are being investigated (e.g. dose level -1) and they have previously tolerated lorlatinib monotherapy at the dose being investigated.
* History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis or pulmonary fibrosis. Patients with history of prior radiation pneumonitis are not excluded.
* Serum albumin ≤ 2.5 g/dL
* History of HIV or history of active tuberculosis
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors, including their administration within 2 weeks prior to the first study treatment (i.e., strong CYP3A4 inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [e.g., Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan; Moderate CYP3A4 inhibitors: erythromycin, verapamil,atazanavir, delavirdine, fluconazole, darunavir, diltiazem, aprepitant, imatinib, tofisopam,ciprofloxacin, cimetidine).
* Current use or anticipated need for drugs that are known strong CYP3A4 inducers including their administration within 2 weeks prior to the first study treatment (i.e., phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St. John's Wort).
* Current symptomatic congestive heart failure or history of symptomatic congestive heart failure in the preceding 3 months, defined as NY Heart Association Classification 2- 4
* Binimetinib and TNO155 groups only: Left ventricular ejection fraction < 50% or institutional lower limit of normal, whichever is lower
* Current diagnosis of symptomatic bradycardia
* Abnormal hematologic and end organ function, defined by the following laboratory results:

  * Absolute neutrophil count ≤ 1500 cells/µL (granulocyte colony-stimulating factor support should not be used within 2 weeks prior to Cycle 1, Day 1).
  * Platelet count ≤100,000/µL
  * Hemoglobin ≤ 9.0 g/dL (patients may be transfused above this threshold)
  * INR and aPTT ≥ 1.5 x ULN. Patients receiving therapeutic anticoagulation may exceed these parameters provided they are on a stable dose.
  * Serum creatinine ≥1.5x the ULN or an estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) equation of < 45 mL/min/1.73 m2
  * Serum lipase ≥ 1.5x ULN
* Liver disease characterized by:

  * ALT or AST ≥ 3x ULN (or > 5x ULN for patients with concurrent liver metastasis)
  * Total bilirubin > 1.5 × ULN; NOTE: Patients with documented Gilbert's syndrome or hyperbilirubinemia due to nonhepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the Overall Principal Investigator.
  * Impaired synthetic function or other conditions of decompensated liver disease, such ascoagulopathy, hepatic encephalopathy, ascites, and bleeding from esophageal varices
  * Acute viral or active autoimmune, alcoholic, or other types of acute hepatitis
* Binimetinib and TNO155 groups only: History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration.
* Major surgical procedure (including brain surgery) within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
* Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, localized/stable renal masses, DCIS/LCIS of the breast, or localized and presumed cured prostate cancer) within the last 3 years.
* Active inflammatory gastrointestinal disease or previous gastric resection or lap band.
* Inability or unwillingness to swallow pills
* Concurrent use of other tyrosine kinase inhibitors
* Prior treatment with a MAP-kinase pathway inhibitor (RAS, RAF, ERK, MEK).
* Allergy or hypersensitivity to components of the lorlatinib, binimetinib, or crizotinibformulations
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would preclude the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose as assessed by CTCAE v5.0. Phase I. | 28 days (binimetinib and crizotinib arm), 21 days (TNO155 arm)
  The highest dose of the combinations that does not cause unacceptable side effects. The maximum tolerated dose is determined in clinical trials by testing increasing doses in different groups of patients until the highest dose with acceptable side effects is found.
The objective response rate, including partial and complete responses, as evaluated by RECIST v1.1. Phase II | 24 months
  Objective response rate (partial and complete responses) will be evaluated according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE V5.0 | From first dose to end of study. Time frame is anticipated to be 24 months.
  Number of patients with treatment-related side effects, according to CTCAE v5.0
Progression-Free Survival as assessed by RECIST v1.1 and the Kaplan-Meier Method | Time from the start of study drug treatment to the date of the first documented progression or death due to disease, likely average of 12 months
  PFS will defined as the time from the start of treatment to the date of the first documented progression or death due to disease. The distribution of PFS will be estimated using the Kaplan-Meier method.
Duration of Response to Treatment as Assessed by RECIST v1.1 | Measured from the time measurement criteria are met for complete or partial response until the first date that recurrent or progressive disease is objectively documented or the date of death due to any cause, likely average of 12 months
  Duration of response to treatment is measured from the time that measurement criteria (RECIST v1.1) are met for complete response or partial response (whichever is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started), or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ibiayi Dagogo-Jack, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team
URL: http://www.partners.org/innovation